CLINICAL TRIAL: NCT06588985
Title: Exploring the Role of Parental Emotion Regulation and Outcomes of Parental Emotional Coaching on Child and Adolescent Psychosocial Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Ministry of Education, Singapore (Other Government)
Responsible Party: Principal Investigator, Ong Jiehan Jamie, Instructor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NUS-IRB-2023-859
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Emotion Regulation
Keywords: Emotion Coaching
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the treatment group or waitlist control group.
Who Masked: Participant
Masking Description: Participants do not know which group they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotion Coaching Treatment Group (Experimental): Parents of the parent-child dyad in this group, will attend 1 3-hour parent workshop on emotion coaching. Followed by 2 biweekly phone consultations with a clinical psychologist.
  Interventions: Behavioral: Emotion Coaching Parent Training Workshop
- Waitlist Control Group (Active Comparator): In this group, questionnaires/data will be collected, but no treatment will be given. Only after they have submitted all data, then they will be invited to participate in the above Emotion Coaching parent workshop and phone consultations.
  Interventions: Behavioral: Waitlist Control

INTERVENTIONS:
Behavioral: Emotion Coaching Parent Training Workshop — Parents will attend a 3-hour online workshop that introduces the fundamentals of emotion coaching and the phone consultations will be used to help parents troubleshoot and brainstorm application of the workshop content.
  Arms: Emotion Coaching Treatment Group
Behavioral: Waitlist Control — Parents will only receive the parent workshop and phone consultations after they have completed all the required questionnaires.
  Arms: Waitlist Control Group

SUMMARY:
Emotional regulation has been found to play a crucial role in an individual's mental well-being and emotional dysregulation is implicated in most of psychiatric disorders listed in the Diagnostic and Statistical Manual, Fifth Edition (DSM-5) (APA, 2013; Gross & Levenson, 1997; Thoits, 1985). Specifically in children, poor emotional regulation skills and parental emotional dysregulation contribute significantly to childhood psychopathology (Han & Shaffer, 2014). This study has two parts - Part 1 aims to explore and identify the parental emotion socialization factors that contributes to a child's emotion regulation abilities and examine how parental emotion dysregulation contribute to the profile of a child's emotional and behavioral difficulties; Part 2 attempts to determine the effectiveness of parental emotional coaching in developing a child's emotion regulation abilities and reducing a child's symptoms of psychopathology. Participants will include both nonclinical and clinical samples, consisting of children and adolescents, aged 7 to 17 years old (middle childhood to adolescence) and their parents. Participants will be invited to complete a set of questionnaires (Part 1) and to participate in a randomized controlled trial that provides parents with a workshop on emotion coaching skills (Part 2). Data will be analysed using correlation,regression analyses and mixed Analysis of Variance (ANOVA). Clinical implications from this study includes, informing of improvements to the clinical services provided in the healthcare setting, as well as contribute to the transdiagnostic formulation of children and adolescent mental health conditions.

DETAILED DESCRIPTION:
Proposed Methodology This research proposes 2 studies to investigate the above stated questions. Study 1 will utilize a cross-sectional design with children and adolescents, as well as their parents (from general population), completing questionnaires provided, while Study 2 will involve inviting participants from Study 1 to participate in a randomized controlled trial. Participants may choose to only participate in Study 1 and not Study 2. If participants are keen and provide consent to participate in Study 2, they will have to complete both interventions and all questionnaires required at all timepoints.

Participants & Procedure Participants include children and adolescents aged 7 to 17 years old, and one of their parents. Participants will be recruited from the community and the Student Health Centre at Health Promotion Board (HPB). HPB is only used as a referral site and recruitment site. Research procedures are not conducted on their premise. Both parents and children will be required to be fluent in the English language, and all parent-child dyads will be invited to participate.

In terms of procedure, interested participants (parent-child dyads) will be invited to participate. Consent will be collected from the child and their parents. For Study 1, after consent is taken, participants will be asked to complete a set of questionnaires and indicate their interest to participate in Study 2. Survey questionnaires will be administered either face-to-face or online - for face-to-face administration, the researcher will provide parent-child dyad with a tablet to complete the questionnaires; for online administration, parent-child dyads will be emailed a link to the questionnaires to complete (most likely on Qualtrics). All participants are advised to complete all questions and do not skip. A copy of the questionnaire will be shown in its entirety to participants before providing consent. For children, if they have difficulty understanding the questions, they are allowed to skip it or seek help from their parents/researcher. The parents' questionnaire should take at most 30 minutes to complete, while the child's questionnaire will take at most 15 minutes to complete.

If participants only participate in Study 1, they will only be required to complete the set of questionnaires at Timepoint 1. Participants in Study 1 will not be debriefed, but they can request to be debriefed by contacting the research team and we can arrange a debrief via Zoom.

In Study 2, a randomized controlled trial is designed to test the effects of parent emotion coaching on parental factors (such as ER skills, sense of competency, and mood and stress levels), child factors (such as ER skills, internalizing and externalizing problems, and treatment outcomes), as well as parent-child relationship. Participants will be a subset of Study 1's participants.

If participants indicate interest to participate in Study 2, the parents will be randomly assigned to the following experimental groups: 1. Emotion Coaching Training, or 2. Waitlist Control condition. Parents in the emotion coaching workshop will be invited to attend an online training on emotion coaching strategies, while parents in the control condition will not be receiving any training workshops during the study. They will be invited to join the online workshops when the study is completed. Participants will not be informed of the group that they are assigned to, and a debrief session will be provided once they complete the study. \

The training module consists of a three-hour workshop, followed by 2 bi-weekly 30-minute phone/online consultations (participants can choose from preferred timeslot on weekdays during regular work hours).

Parents and children will be required to complete the set of outcome measures at pre-, post-treatment and at a 1-month follow-up. All procedures are conducted in English only.

Estimated timeline for the different groups:

Treatment Group - Week 0: Questionnaire (parent and child), Weeks 1 - 5: Parent Workshop, 2 phone consults, Week 6: post-questionnaire (parent and child), Week 9 - 10: follow-up questionnaire (parent and child). Intervention phase itself will last at most 5 weeks. The 3-hour online workshop will be conducted in real-time over Zoom, by a clinical psychologist or a Masters in Clinical Psychologist student (supervised by a clinical psychologist).

Waitlist Group - Week 0: Questionnaire (parent and child), Week 6: Questionnaire T2 (parent and child), Week 9-10: Questionnaire T3 (parent and child). After they have completed all 3 sets of questionnaires, they will be invited to sign up for the workshop on dates that are convenient for them. The 3-hour online workshop will be conducted in real-time over Zoom, by a clinical psychologist or a Masters in Clinical Psychologist student (supervised by a clinical psychologist).

At the end of Study 2, all participants will be provided with the debrief sheet (either hard or soft copy can be provided) and offered a debrief session over Zoom. The debrief session will be conducted by the research team.

In cases whereby participants may wish to have longer consultation sessions, or to extend the intervention outside of the research, they may be referred to the relevant professionals/services.

Participants have until 1 week after they completed the study to decide if they wish to withdraw their research data.

ELIGIBILITY:
Inclusion Criteria:

* Participants include children and adolescents aged 7 to 17 years old, and one of their parents.
* All parent-child dyads will be invited to participate.
* Parents and children have to be fluent in English.
* Persons who are not parents will not be recruited.

Exclusion Criteria:

* Children or parents with physical impairments (apart from corrected vision) will be excluded.
* Children or parents reporting psychotic symptoms, neurodevelopmental disorders, or severe mood disorders will be excluded.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-05-24 (Estimated); Study Completion 2026-05-24 (Estimated)

PRIMARY OUTCOMES:
Emotion Regulation Questionnaire (ERQ; Gross & John, 2003) | Baseline, 1-month after baseline and at least 2-months after baseline
  ERQ is a self-report questionnaire designed to measure an individual's tendency to regulate their emotions in 2 ways: cognitive reappraisal and expressive suppression. There are 10 items, and each item is rated on a 7-point Likert scale of 1 (Strongly Disagree) to 7 (Strongly Agree). The scores of each scale will be calculated separately and the higher a score on a scale indicates higher tendency for the individual to use the specific method to regulate their emotions.
Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA; Gullone & Taffe, 2011) | Baseline, 1-month after baseline and at least 2-months after baseline
  ERQ-CA is adapted from the ERQ for adults to be used to measure a child's tendency to regulate their emotions on the 2 scales: cognitive reappraisal and expressive suppression. Similar to the ERQ, it has 10 items rated on a 7-point Likert Scale (from 1 (Strongly Disagree) to 7 (Strongly Agree)). Higher scores on each scale indicates higher tendency to use the corresponding method to regulate their emotions. The ERQ-CA demonstrated sound internal consistency, as well as sound construct and convergent validity (Gullone & Taffe, 2011).
Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) | Baseline, 1-month after baseline and at least 2-months after baseline
  DERS is a 36-item self-report questionnaire that measure the types of emotion regulation and dysregulation an individual might experience. Items are rated on a 5-point Likert scale, ranging from 1 (Almost Never) to 5 (Almost Always). The items measure how often the individual might engage in each of the behaviours or have specific thoughts. The items can be grouped into 6 subscales: nonacceptance of emotional responses, difficulty engaging in goal-directed behaviour, impulse control difficulties, lack of emotional awareness, limited access to emotional regulation strategies, and lack of emotional clarity. The scores are added up and higher scores indicate greater problems with emotion regulation. The DERS was found to have good internal consistency, test-retest reliability and adequate construct and predictive validity (Gratz & Roemer, 2004).

SECONDARY OUTCOMES:
Depression Anxiety Stress Scales short version (DASS-21; Lovibond & Lovibond, 1995) | Baseline, 1-month after baseline and at least 2-months after baseline
  DASS 21 is a 21-item self-report scale that measures an individual's negative emotional states of depression, anxiety and stress. Each item has 4 options ranging from 0 (did not apply to me at all) to 3 (applied to me much, or most of the time). Higher scores on each scale indicates elevated symptoms of depression, anxiety and stress respectively. The DASS-21 have shown good reliability and validity (Lovibond & Lovibond, 1995).
Parent Sense of Competency (PSOC; Gilmore & Cuskelly, 2008) | Baseline, 1-month after baseline and at least 2-months after baseline
  PSOC is a 17-item self-report questionnaire that measure parents' satisfaction with parenting and their self-efficacy in the parenting role. The items are rated on a 6-point Likert Scale (from 1 (Strong Disagree) to 6 (Strongly Agree)). The scores are added up, and a higher score indicates a higher parental sense of competency. Good internal consistency and validity were demonstrated (Gilmore & Cuskelly, 2008).
Parent Relationship Questionnaire (PRQ; Kamphaus & Reynolds, 2006) | Baseline, 1-month after baseline and at least 2-months after baseline
  PRQ is a 71-item questionnaire that assesses parents' perceptions of attachment, communication, discipline, involvement, confidence, satisfaction with child's school, and relational frustration. Each item is rated on a 4-point Likert scale (N = Never, S = Sometimes, O = Often, and A = Always). Parents will be asked to circle the best answer that represents their beliefs about or experiences with their child. Scores are presented in the form of T-scores. Lower scores on the Attachment, Communication, Discipline Practices, Involvement, Parenting Confidence, and Satisfaction with School scale, indicates more relationship problems. In contrast, higher scores on the Relational Frustration scale indicates more problems. PRQ was found to have good internal consistency and adequate validity (Rubinic & Schwickrath, 2010).
Security Scale questionnaire (SSQ; Kerns et al., 1996) | BBaseline, 1-month after baseline and at least 2-months after baseline
  The SSQ consists of 15-items evaluating children's view of attachment security with a particular attachment figure (e.g. mother). It employs the "Some kids. . . Other kids. . ." structure pioneered by Susan Harter (1982). For example, "Some kids are more confident trying new things after talking to their mom about it, BUT other kids do not feel more confident trying new things after talking to their mom about it". The scoring takes the summation of all items to obtain a single score on a security dimension, with higher scores indicating greater security. The scale demonstrated sound reliability and validity with alphas of .84 and .88, respectively (Kerns et al., 1996).
Big-Five Questionnaire for Children (BFQ-C; Barbaranelli et al., 2003) | Baseline only
  The BFQ-C consists of 65-items measuring the five personality factors in children: 1) openness/intellect, 2) conscientiousness, 3) extraversion/energy, 4) agreeableness, and 5) neuroticism/emotional instability. Items are rated on a 5-point Likert scale varying from 1 (almost never) to 5 (almost always). The scoring takes the summation of all items in each of the five factors, with a higher score on each factor indicating a higher score for that particular personality trait. The subscales demonstrated good internal consistency (Cronbach's alpha = .80 - .99) (Barbaranelli et al., 2003).

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ong, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT06588985/Prot_000.pdf
  • Informed Consent Form (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT06588985/ICF_001.pdf